CLINICAL TRIAL: NCT04614012
Title: The Use of Hyperimmune Plasma for the Treatment of COVID-19 Infection
Brief Title: Hyperimmune Plasma for Patients With COVID-19
Acronym: IMMUNO-COVID19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANNA FALANGA (Other)
Responsible Party: Sponsor-Investigator, ANNA FALANGA, Prof, A.O. Ospedale Papa Giovanni XXIII
Organization: A.O. Ospedale Papa Giovanni XXIII (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMUNO-COVID19
Record Dates: First submitted 2020-11-02; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: covid19; Hospitalized patients; Hyperimmune plasma
MeSH Terms: conditions — COVID-19 | interventions — Therapeutics; COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Longitudinal assessment of COVID-19 patients treated with hyperimmune plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hyperimmune plasma (Experimental): treated with hyperimmune plasma
  Interventions: Other: treated with hyperimmune plasma

INTERVENTIONS:
Other: treated with hyperimmune plasma — administration of hyperimmune plasma at day 1 and based on clinical response on day 3 and 5
  Other Names: hyperimmune plasma

SUMMARY:
The outbreak of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which originated in Wuhan, China, has become a major concern all over the world.

Convalescent plasma or immunoglobulins have been used as a last resort to improve the survival rate of patients with SARS whose condition continued to deteriorate despite treatment with pulsed methylprednisolone. Moreover, several studies showed a shorter hospital stay and lower mortality in patients treated with convalescent plasma than those who were not treated with convalescent plasma. Evidence shows that convalescent plasma from patients who have recovered from viral infections can be used effectively as a treatment of patients with active disease. To date, no specific treatment has been proven to be effective. The investigators plan to treat critical Covid-19 patients with hyperimmune plasma.

DETAILED DESCRIPTION:
Apheresis from recovered donors will be performed with a cell separator device , with 500-600 mL of plasma obtained from each donor. Donors are males and womens , age 18 yrs or more, evaluated for transmissible diseases according to the italian law. Adjunctive tests will be for hepatitis A virus, hepatitis E virus and Parvovirus B-19. All donors will be tested for the Covid-19 neutralizing title. Each plasma bag obtained from plasmapheresis will be immediately divided in two units and frozen according to the national standards and stored separately.

Based on experience published in literature 250-300 mL of convalescent plasma will be used to treat each of the recruited patients at most 3 times over 5 days.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 yrs
* positive for reverse transcription polymerase chain reaction (RT-PCR) severe acute respiratory syndrome (SARS)-CoV-2
* Acute respiratory distress syndrome (ARDS) moderate to severe, according to Berlin definition, lasting less than10 days
* Polymerase chain reaction (PCR) positive
* signed informed consent unless unfeasible for the critical condition

Exclusion Criteria:

* proven hypersensitivity or allergic reaction to hemoderivatives or immunoglobulins
* consent denied

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-07-02 (Estimated); Study Completion 2022-07-02 (Estimated)

PRIMARY OUTCOMES:
Death | within 30 days
  death from any cause

SECONDARY OUTCOMES:
time to extubation | within 7 days
  days since intubation
length of intensive care unit stay | within 7 days
  days from entry to exit from ICU
length of hospitalization | within 30 days
  days from entry to exit from hospital
immune response | at days 1, 3 and 7
  neutralizing title
viral load | at days 1, 3 and 7
  naso-pharyngeal swab and BAL

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Falanga, Bergamo, Italy